CLINICAL TRIAL: NCT06070883
Title: Efficacy of Mutilayered Fresh Amnoitic Membrane Transplantation in Resistant Fungal Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Resistant fungal keratitis
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amniotic membrane (Other): Amniotic membrane (AM) is the innermost layer of the placenta, which consists of a single layer of meta-bolically active epithelium, a thick basement membrane, and an avascular stromal matrix.It has been shown to exhibit a wide array of biological properties, including wound healing, anti-inflammatory, antimicrobial, and anti-angiogenic properties, amongst others
  Interventions: Procedure: Amniotic membrane transplantation

INTERVENTIONS:
Procedure: Amniotic membrane transplantation — Amniotic membrane (AM) is the innermost layer of the placenta, which consists of a single layer of meta-bolically active epithelium, a thick basement membrane, and an avascular stromal matrix. It has been shown to exhibit a wide array of biological properties, including wound healing, anti-inflammatory, antimicrobial, and anti-angiogenic properties, amongst others. Amniotic membrane transplantation will be performed in eye OT under aseptic conditions. The necrotic tissues at the base of the ulcer will be debrided and sent for culture and sensitivity. The rolledup edge of the ulcer or the loosely adhered epithelium adjacent to the ulcer will also be removed. The amniotic membrane will be trimmed to fit the shape of the ulcer and placed with its epithelial side up. Then the amniotic membrane will be secured with 10-0 nylon suture (5 cases with interrupted and 25 cases with continuous suture) with the suture knots buried.

SUMMARY:
Corneal infection or infectious keratitis (IK) is the most common cause of corneal blindness worldwide, particu-larly in the developing countries1. The incidence was estimated at 2.5-799 per 100,000 population/year. It is a painful and potentially blinding ocular emergency that often requires hospital admission for intensive medical and/or surgical treatment. Depending on the geographical and temporal variations and population-based risk factors (e.g. agricultural practice, trauma, use of contact lens and others), bacteria and fungi have been shown to be the main causative microorganisms for IK, followed by viruses, parasites and polymicrobial infection. Amniotic membrane (AM) is the innermost layer of the placenta, which consists of a single layer of meta-bolically active epithelium, a thick basement membrane, and an avascular stromal matrix (15).

It has been shown to exhibit a wide array of biological properties, including wound healing, anti-inflammatory, antimicrobial, and anti-angiogenic properties, amongst others. To date, a number of studies have evaluated the benefit of AMT for treating active IK, though the majority of them were of small case series or case reports. In clinical practice, AMT is usually reserved as a second-line therapy in IK, mainly to promote cornea healing in non-healing ulcer after the sterilization phase.

ELIGIBILITY:
Inclusion Criteria:

* Size more than 5 mm.
* Deep ulcers i.e. > 50% stromal thickness.
* Located within 3mm of the visual axis.
* Patients with descemetoceles and corneal perforations will also be included

Exclusion Criteria:

* Corneal ulcers of size < 5mm depth < 50%
* Associated glaucoma
* Associated chronic dacryocystitis
* Ulcers with entropion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Corneal Pain | Baseline
  it will be meaured by the Visual analouge scale
Corneal Pain | one month post operative
  it will be meaured by the Visual analouge scale
Corneal Pain | three months post operative
  it will be meaured by the Visual analouge scale
Size of the ulcer | Baseline
  it will be meaured in mellimeter
Size of the ulcer | one month post operative
  it will be meaured in mellimeter
Size of the ulcer | three months post operative
  it will be meaured in mellimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No